CLINICAL TRIAL: NCT04798781
Title: A Phase II Study Evaluating Safety and Efficacy of Telatinib in Combination With Keytruda in Subjects With Advanced Stomach and Gastroesophageal Junction Cancers or Hepatocellular Carcinoma
Brief Title: Safety and Efficacy of Telatinib in Combination With Keytruda in Subjects With Advanced Stomach and Gastroesophageal Junction Cancers or Hepatocellular Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Andrew Hendifar, MD (Other)
Collaborators: EOC Pharma (Industry)
Responsible Party: Sponsor-Investigator, Andrew Hendifar, MD, Assistant Professor, Medicine, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2020-11-Hendifar-TELAT
Record Dates: First submitted 2021-02-24; First posted 2021-03-15 (Actual); Results first posted 2024-10-10 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Gastric Cancer; Hepatocellular Carcinoma
MeSH Terms: conditions — Stomach Neoplasms; Carcinoma, Hepatocellular | interventions — telatinib; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- telatinib + Keytruda (Experimental)
  Interventions: Drug: Telatinib; Drug: Keytruda

INTERVENTIONS:
Drug: Telatinib — 900mg by mouth twice daily until disease progression, intolerable toxicities, or withdrawal of consent
Drug: Keytruda — 200mg intravenous infusion every three weeks until disease progression, intolerable toxicities, or withdrawal of consent
  Other Names: pembrolizumab

SUMMARY:
This is a phase II, single arm, open-label study of two parallel cohorts (advanced stomach and gastroesophageal junction cancer and hepatocellular carcinoma), evaluating the effects of telatinib in combination with Keytruda on progression-free survival.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: Histologically confirmed gastric/esophagealgastric adenocarcinoma, recurrent, locally advanced or metastatic, PD-L1-positive disease (CPS ≥1), progressed on at least two prior lines of therapy and/or discontinued second line therapy for intolerance, indicated for Keytruda therapy. OR: Hepatocellular carcinoma with diagnosis confirmed by histologic or cytologic analysis or clinical features according to the American Association for the Study of Liver Diseases criteria for patients with cirrhosis, unresectable disease not amenable to locoregional therapy with disease progression after at least one prior line of systemic therapy or discontinued first line therapy for intolerance.
* At least 1 measurable metastatic lesion that has not been irradiated. The lesion will be measured according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1), and be documented by radiological evaluation within 28 days prior to registration. For subjects with locally advanced disease: at least one measurable lesion that has not been irradiated, documented by radiological evaluation within 28 days prior to registration.
* Any prior radiation therapy must be completed at least 28 days prior to the first dose of study treatment.
* Eighteen years of age or older.
* Eastern Cooperative Oncology Group (ECOG) performance score of 0, 1 or 2.
* Adequate bone marrow, liver, and renal function
* Negative urine or serum pregnancy test for women of childbearing potential.
* Women and men of childbearing potential must agree to use adequate contraception prior to registration, for the duration of study participation and until 4 months after the last study drug dosing.
* Able to swallow tablets and agree to take the prescribed tablets twice daily.

Exclusion Criteria:

* Clinical or radiographic evidence of current brain metastasis. History of treated brain metastases is allowable.
* Cardiac disease
* Uncontrolled hypertension
* Severe hemorrhage/bleeding event within 28 days prior to the first dose of study treatment
* Major surgery, open biopsy, or significant traumatic injury within 42 days prior to the first dose of study treatment
* Current serious, nonhealing wound, ulcer, or bone fracture within 42 days prior to the first dose of study treatment
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to the first dose of study treatment.
* Presence of an uncontrolled infection or infection that required intravenous antibiotics, antifungals, or antivirals within 14 days prior to the first dose of study treatment.
* Known human immunodeficiency virus (HIV) infection. HIV-infected subjects on effective anti-retroviral therapy are eligible if the most recent viral load test performed within six months of screening (based on medical chart review) is negative. The safety of telatinib in this subject population has not been studied.
* Known chronic hepatitis B, unless receiving antiviral treatment.
* Known Child-Pugh Score B or C liver cirrhosis.
* Diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment or has been diagnosed with an autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs). Patients that require replacement therapy (e.g., thyroxine [T4], insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) may be enrolled.
* History of (non-infectious) pneumonitis that required steroids, or current pneumonitis, or has a history of interstitial lung disease.
* Has received a live-virus vaccination within 30 days of planned treatment start.
* Known history of proteinuria > 1gr/24 hours.
* Previous or concurrent cancer that is distinct in primary site or histology from the current stomach or liver cancer. Subjects with cervical cancer in-situ, treated basal cell carcinoma, superficial bladder tumors (Ta and Tis) or any cancer curatively treated are not excluded.
* Anti-cancer therapy (chemotherapy, hormonal therapy, radiation therapy, surgery, immunotherapy, biologic therapy, or tumor embolization) or investigational agent within 28 days prior to the first dose of study treatment.
* Known or suspected allergy to any component of telatinib or Keytruda
* Prior or current history of substance abuse, or medical, psychological, or social condition that in the opinion of the investigator may interfere with the subject's participation in the study or evaluation of the study result.
* Women who are pregnant or breastfeeding.
* Prior history of thromboembolic disease, e.g., deep vein thrombosis (DVT), pulmonary emboli (PE), within 6 months prior to the first dose of study treatment that has required continued medical intervention.
* Baseline peripheral neuropathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-07-28 (Actual); Primary Completion 2024-02-14 (Actual); Study Completion 2025-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Hendifar, MD, MPH, Principal Investigator — Cedars-Sinai Medical Center
Locations (3):
- United States (3):
  - CS Cancer Beverly Hills, Beverly Hills, California
  - CS Cancer at The Angeles Clinic and Research Institute, Los Angeles, California
  - CS Cancer at the Samuel Oschin Cancer Center, Los Angeles, California

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial opened to accrual on 7/12/2021 with first subject enrolled on study 7/28/2021. A total of 23 patients consented; 5 subjects failed screening; 2 were withdrawn; 16 subjects went on treatment, 1 subject (subject 009) withdrew consent; 15 completed study intervention evaluable. The study was closed to accrual on 02/07/2023 due to discontinuation of support by the drug supplier and funding source, due to postulated limited potential utility of the study drug.
Groups:
- telatinib + Keytruda: Telatinib: 900mg by mouth twice daily until disease progression, intolerable toxicities, or withdrawal of consent
  Keytruda: 200mg intravenous infusion every three weeks until disease progression, intolerable toxicities, or withdrawal of consent
  Single Arm with 2 Cohorts:
  Cohort 1: Gastric/esophagealgastric adenocarcinoma, recurrent, locally advanced or metastatic, PD-L1-positive disease (CPS ≥1), progressed on at least two prior lines of therapy and/or discontinued second line therapy for intolerance, indicated for Keytruda therapy.
  Cohort 2: Hepatocellular carcinoma, with diagnosis confirmed by histologic or cytologic analysis or clinical features according to the American Association for the Study of Liver Diseases criteria for patients with cirrhosis, unresectable disease not amenable to locoregional therapy with disease progression after at least one prior line of systemic therapy or discontinued first line therapy for intolerance.
Period: Overall Study
Arm/Group | telatinib + Keytruda
Started | 16
Completed | 15
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Telatinib + Keytruda
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.93 (14.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Duration of time from start of treatment until progression or death, whichever comes first
Time Frame: through study completion, approximately 2.5 years
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | telatinib + Keytruda
Number analyzed (Participants) | 15
Days | 153.87 (133.69)

2. Secondary Outcome: Overall Response Rate
Description: The percentage of patients who have a partial or complete response to treatment
Time Frame: from the start of treatment until the end of treatment, approximately 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | telatinib + Keytruda
Number analyzed (Participants) | 15
Participants | 0

3. Secondary Outcome: Disease Control Rate
Description: The percentage of patients who have stable disease, partial response, or complete response to treatment
Time Frame: from the start of treatment until the end of treatment, approximately 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | telatinib + Keytruda
Number analyzed (Participants) | 15
Participants | 8

4. Secondary Outcome: Overall Survival
Description: The length of time from the start of treatment that patients are still alive
Time Frame: from the start of treatment until time-of-event
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | telatinib + Keytruda
Number analyzed (Participants) | 15
days | 258 [116 to 1238]

5. Secondary Outcome: Number and Severity of Adverse Events
Description: Incidence and severity of adverse events as measured by the National Cancer Institute Common Terminology Criteria for Adverse Events Version 5
Time Frame: from the start of treatment until 30 days following the end of treatment or until initiation of a new anticancer therapy (whichever occurs first), approximately 13 months
Measure: Count of Units; unit: Adverse Events (AEs)
Units Other Than Participants: Adverse Events (AEs)
Arm/Group | telatinib + Keytruda
Number analyzed (Participants) | 16
Number analyzed (Adverse Events (AEs)) | 313
Adverse Events (AEs)
  Grade 1 | 161
  Grade 2 | 87
  Grade 3 | 57
  Grade 4 | 7
  Grade 5 | 1

ADVERSE EVENTS:
Time Frame: approximately 13 months
Description: All patients experiencing an AE will be monitored until: the AE resolves or the symptoms or signs that constitute the AE return to baseline, any abnormal laboratory value deemed an AE, has returned to baseline, there is a satisfactory explanation other than the study drug for the changes observed, death, or until 30 days following last dose of study drug or until initiation of a new anticancer therapy (whichever occurs first)
Arm/Group | telatinib + Keytruda
All-Cause Mortality (participants affected / at risk) | 12/16
Serious Adverse Events (participants affected / at risk) | 8/16
Other Adverse Events (participants affected / at risk) | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | telatinib + Keytruda (N=16)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Biliary tract infection (Infections and infestations) | 1 (4)
Blood Bilirubin Increased (Investigations) | 1 (3)
Constipation (Gastrointestinal disorders) | 1 (3)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Hepatic Failure (Hepatobiliary disorders) | 3 (7)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2)
Lung Infection (Infections and infestations) | 1 (2)
Other (Metabolism and nutrition disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | telatinib + Keytruda (N=16)
Abdominal pain (Gastrointestinal disorders) | 3 (5)
Alanine Aminotransferase (Investigations) | 5 (16)
Alkaline Phosphatase Increased (Investigations) | 1 (5)
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Anal Fistula (Gastrointestinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 5 (17)
Anorexia (Metabolism and nutrition disorders) | 3 (4)
Anxiety (Psychiatric disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (4)
Ascites (Gastrointestinal disorders) | 3 (3)
Asparate Aminotransferase Increased (Investigations) | 5 (17)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Blood Bilirubin Increased (Investigations) | 4 (10)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Buttock Pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Chest Pain- Cardiac (Cardiac disorders) | 1 (1)
Chills (General disorders) | 1 (2)
Conjunctivitis (Infections and infestations) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Creatinine Increased (Investigations) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 6 (10)
Dizziness (Nervous system disorders) | 2 (3)
Dry Mouth (Gastrointestinal disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Dyspnea (Renal and urinary disorders) | 2 (2)
Dysuria (Renal and urinary disorders) | 1 (2)
Edema Face (General disorders) | 1 (1)
Edema Limbs (General disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Eye Disorders- Other, Specify (Eye disorders) | 1 (1)
Eye Pain (Eye disorders) | 1 (1)
Facial Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (2)
Fatigue (General disorders) | 10 (19)
Fever (General disorders) | 1 (1)
Gait Disturbance (General disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (3)
General Disorders and Administration Site Conditions - Other, Specify (General disorders) | 1 (1)
General Disorders and Administration Site Conditions - Other, Specify (Gastrointestinal disorders) | 1 (1)
Generalized Edema (General disorders) | 1 (1)
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 3 (3)
Genital Edema (Reproductive system and breast disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Hepatic Failure (Hepatobiliary disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hip Fracture (Injury, poisoning and procedural complications) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 3 (20)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 2 (2)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Localized Edema (General disorders) | 1 (1)
Mucositis Oral (Gastrointestinal disorders) | 2 (2)
Muscle Cramp (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - other, specify (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (6)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 9 (10)
Nausea (Investigations) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neutrophil Count Decreased (Investigations) | 1 (1)
Other (Musculoskeletal and connective tissue disorders) | 1 (1)
Other (Eye disorders) | 1 (1)
Other (Investigations) | 1 (1)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Papulopustular Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Pelvic Pain (Reproductive system and breast disorders) | 1 (1)
Periorbital Edema (Eye disorders) | 1 (1)
Platelet Count Decreased (Investigations) | 4 (8)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2)
Rash Acneiform (Skin and subcutaneous tissue disorders) | 2 (5)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 2 (2)
Rectal Fissure (Gastrointestinal disorders) | 1 (2)
Rectal Pain (Gastrointestinal disorders) | 1 (1)
Renal and Urinary Disorders - Other, specify (Renal and urinary disorders) | 1 (2)
Skin Infection (Skin and subcutaneous tissue disorders) | 1 (1)
Skin Infection (Infections and infestations) | 1 (1)
Sleep Apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Stomach Pain (Gastrointestinal disorders) | 2 (3)
Thrush (Infections and infestations) | 1 (1)
Upper Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 1 (1)
Urinary Frequency (Renal and urinary disorders) | 2 (2)
Urinary Tract Infection (Infections and infestations) | 3 (5)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1)
Vaginal Infection (Infections and infestations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 6 (8)
Weight Loss (Investigations) | 5 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-15): https://cdn.clinicaltrials.gov/large-docs/81/NCT04798781/Prot_SAP_000.pdf
  • Informed Consent Form (2021-10-26): https://cdn.clinicaltrials.gov/large-docs/81/NCT04798781/ICF_001.pdf